CLINICAL TRIAL: NCT02981069
Title: Effect of Chronic Exenatide Therapy on Beta Cell Function and Insulin Sensitivity in Type 2 Diabetes Mellitus (T2DM)
Brief Title: Effect of Chronic Exenatide Therapy on Beta Cell Function and Insulin Sensitivity in T2DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20160597H
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Byetta / Bydureon (Active Comparator): Exenatide:
  4 weeks Byetta, 5 to 10ug sc (daily) 12 weeks Bydureon 2mg sc
  Interventions: Drug: Exenatide
- Dapagliflozin (Active Comparator): 4 weeks Dapagliflozin, Farxiga, 10mg 12 weeks Dapagliflozin, Farxiga, 10mg
  Interventions: Drug: Dapagliflozin
- Byetta/Bydureon plus Dapagliflozin (Active Comparator): Exenatide:
  4 weeks Byetta, 5 to 10ug sc (daily) 12 weeks Bydureon 2mg sc PLUS
  Dapagliflozin:
  4 weeks Dapagliflozin, Farxiga, 10mg 12 weeks Dapagliflozin, Farxiga, 10mg
  Interventions: Drug: Dapagliflozin; Drug: Exenatide
- Placebo (Placebo Comparator): Placebo group (4 weeks and 12 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10mg
  Other Names: Farxiga
  Arms: Byetta/Bydureon plus Dapagliflozin; Dapagliflozin
Drug: Exenatide — Byetta 5 to 10 ug (twice daily) Bydureon 2mg (once weekly)
  Other Names: Byetta, Bydureon
  Arms: Byetta / Bydureon; Byetta/Bydureon plus Dapagliflozin
Drug: Placebo — Placebo for Dapagliflozin
  Arms: Placebo

SUMMARY:
In this study, the researchers hope to learn about SGLT2 inhibition on EGP (endogenous glucose production) and plasma glucose concentration in diabetic subjects. Researchers will examine diabetes and the role of increased plasma glucagon, decline in plasma insulin, and fall in plasma glucose concentration.

DETAILED DESCRIPTION:
This study will examine whether the coadministration of exenatide plus dapagliflozin will prevent the increase in EGP and result in an additive or even synergistic decrease in plasma glucose concentration compared to each agent alone.

ELIGIBILITY:
Inclusion Criteria:

1. BMI = 25-35 kg/m^2
2. must be drug naïve and/or on a stable dose (more than 3 months) of metformin and/or sulfonylurea
3. HbA1c >7.0% and <10.0%
4. Other than diabetes, subjects must be in good general health as determined by physical exam, medical history, blood chemistries, CBC, TSH, T4, EKG and urinanalysis.
5. Only subjects whose body weight has been stable (± 3 lbs) over the preceding three months and who do not participate in an excessively heavy exercise program will be included.

Exclusion Criteria:

1. Presence of significant systemic disease, heart problems including congestive heart failure, unstable angina or acute myocardial infarction, current infectious liver disease, acute stroke or transient ischemic attacks, history of pancreatitis, urosepsis and pyelonephritis, genital mycotic infections, or Type 1 diabetes mellitus
2. Any hepatic diseases in the past (infectious liver disease, viral hepatitis, toxic hepatic damage, jaundice of unknown etiology) or severe hepatic insufficiency and/or significant abnormal liver function tests defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN
3. Renal impairment (e.g., serum creatinine levels ≥1.4 mg/dL for women or ≥1.5 mg/dl for men, or eGFR <60 mL/min/1.73 m2) or history of unstable or rapidly progressing renal disease or end stage renal disease.
4. Uncontrolled thyroid disease , Cushing's syndrome, congenital adrenal hyperplasia or hyperprolactinemia
5. Significantly elevated triglyceride levels (fasting triglyceride > 400 mg/dl), uncontrolled increased LDL-C
6. Untreated or poorly controlled hypertension (sitting blood pressure > 160/95 mm Hg)
7. Use of anti-obesity drugs or weight loss medications (prescription or OTC) and medications known to exacerbate glucose tolerance (such as isotretinoin, , GnRH agonists, glucocorticoids, anabolic steroids, C-19 progestins) stopped for at least 8 weeks. Use of anti-androgens that act peripherally to reduce hirsutism such as 5-alpha reductase inhibitors (finesteride, spironolactone, flutamide) stopped for at least 4 weeks
8. Prior history of a malignant disease requiring chemotherapy, prior history of bladder cancer regardless treatment
9. Patients at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics should have careful monitoring of their volume status
10. History of unexplained microscopic or gross hematuria, or microscopic hematuria at visit 1, confirmed by a follow-up sample at next scheduled visit.
11. Presence of hypersensitivity to dapagliflozin or other SGLT2 inhibitors (e.g. anaphylaxis, angioedema, exfoliative skin conditions
12. Known hypersensitivity or contraindications to use GLP1 receptor agonists (exenatide, liraglutide)
13. Use of , thiazolidinediones, GLP-1 receptor agonists, DPP-4 inhibitors, SGLT2 inhibitors stopped for at least 8 weeks.
14. Eating disorders (anorexia, bulimia) or gastrointestinal disorders
15. Suspected pregnancy (documented negative serum β-hCG test), desiring pregnancy in next 6 months, breastfeeding, or known pregnancy in last 2 months
16. Active history of illicit substance abuse or significant intake of alcohol
17. Having a history of bariatric surgery
18. Patient not willing to use two barrier method contraception during study period (unless sterilized or have an IUD)
19. Debilitating uncontrolled psychiatric disorder such as psychosis or neurological condition that might confound outcome variables
20. Inability or refusal to comply with protocol
21. Current participation or participation in an experimental drug study in previous three months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2023-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Cersosimo, MD,PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Type 2 diabetes with significant clinical complications were excluded
Groups:
- Byetta / Bydureon: Exenatide:
  4 weeks Byetta, 5 to 10ug sc (daily) 12 weeks Bydureon 2mg sc
  Exenatide: Byetta 5 to 10 ug (twice daily) Bydureon 2mg (once weekly)
- Byetta/Bydureon Plus Dapagliflozin: Exenatide:
  4 weeks Byetta, 5 to 10ug sc (daily) 12 weeks Bydureon 2mg sc PLUS
  Dapagliflozin:
  4 weeks Dapagliflozin, Farxiga, 10mg 12 weeks Dapagliflozin, Farxiga, 10mg
  Dapagliflozin: 10mg
  Exenatide: Byetta 5 to 10 ug (twice daily) Bydureon 2mg (once weekly)
Period: Acute Portion of Study
Arm/Group | Byetta / Bydureon | Dapagliflozin | Byetta/Bydureon Plus Dapagliflozin | Placebo
Started | 25 | 25 | 25 | 15
Completed | 25 | 25 | 25 | 15
Not Completed | 0 | 0 | 0 | 0
Period: 16 Week Drug Administration Period
Arm/Group | Byetta / Bydureon | Dapagliflozin | Byetta/Bydureon Plus Dapagliflozin | Placebo
Started (Since subjects are Type 2 diabetics, there was no placebo arm for this portion of the study. Only 3 arms of the study were conducted: (i) Byetta/Bydureon, (ii) Dapagliflozin (iii) Byetta/Bydureon plus Dapagliflozin.) | 25 | 25 | 25 | 0
Completed | 25 | 25 | 25 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Byetta / Bydureon | Dapagliflozin | Byetta/Bydureon Plus Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 25 | 15 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 23 | 14 | 87
  >=65 years | 0 | 0 | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (3) | 51 (2) | 49 (4) | 54 (3) | 52 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 16 | 8 | 51
  Male | 10 | 13 | 9 | 7 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 19 | 21 | 11 | 67
  Not Hispanic or Latino | 9 | 6 | 3 | 2 | 20
  Unknown or Not Reported | 0 | 0 | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 7 | 6 | 5 | 26
  White | 17 | 17 | 19 | 8 | 61
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 25 | 15 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change in Endogenous Glucose Production (EGP) After Acute Exposure to a Single Dose and Again After 16 Weeks of Treatment
Description: After screening, eligible subjects will receive a measurement of endogenous glucose production (EGP) with a prime-continuous infusion of 3-3H-glucose. The EGP measurement will be performed in the morning after a 10-12 hour overnight fast and will last 8.5 hours (from 6 AM to 2:30 PM). After a 3.5-hour tracer equilibration period, subjects (20 per group) will receive one of the following medications: (i) placebo; (ii) exenatide 5 ug subcutaneously; (iii) dapagliflozin (10 mg); and (iv) dapagliflozin 10 mg + exenatide 5 ug [ACUTE STUDY].
Time Frame: ACUTE [after a single dose of each study drug or placebo]
Population: Type 2 diabetes
Measure: Mean (Standard Error); unit: mg/kg.min
Groups:
- EXENATIDE: Exenatide:
  After acute exposure to a single dose of Exenatide, 5 mcg.
- Dapagliflozin: After acute single dose exposure of Dapagliflozin, Farxiga, 10mg
- Exenatide Plus Dapagliflozin: After acute exposure to both dapagliflozin, farxiga 10 mg orally and a single subcutaneous injection of Exenatide
- Placebo: After a single dose of placebo
Arm/Group | EXENATIDE | Dapagliflozin | Exenatide Plus Dapagliflozin | Placebo
Number analyzed (Participants) | 25 | 25 | 25 | 15
mg/kg.min | -0.18 (0.02) | 0.14 (0.03) | -0.08 (0.03) | -0.03 (0.02)

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) Concentration
Description: The change in (FPG) above baseline following administration of study interventions after 16 weeks of treatment with each study drug(s) compared to data obtained during the acute exposure. Placebo arm was not included in this 16 week portion of the study, since subjects are diabetic. Only 3 arms of the study were conducted: (i) Byetta/Bydureon, (ii) Dapagliflozin (iii) Byetta/Bydureon plus Dapagliflozin.
Time Frame: 16 weeks
Population: type 2 diabetes
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Byetta / Bydureon | Dapagliflozin | Byetta/Bydureon Plus Dapagliflozin
Number analyzed (Participants) | 25 | 25 | 25
mg/dl | 42 (1) | 72 (3) | 11 (3)

3. Secondary Outcome: Change in Plasma Glucagon Concentration
Description: Measurement of change in plasma glucagon concentration after 16 weeks of treatment with each study drug(s) compared to acute exposure at baseline. Placebo arm was not included in this 16 week portion of the study, since subjects are diabetic. Only 3 arms of the study were conducted: (i) Byetta/Bydureon, (ii) Dapagliflozin (iii) Byetta/Bydureon plus Dapagliflozin.
Time Frame: Baseline to 16 weeks
Population: type 2 diabetes
Measure: Mean (Standard Error); unit: pg/ml
Groups:
- Dapa+Exe: Combination dapagliflozin plus exenatide therapy
- Dapa: Dapagliflozin therapy for 16 weeks
- Exenatide: Exenatide therapy for 16 weeks
Arm/Group | Dapa+Exe | Dapa | Exenatide
Number analyzed (Participants) | 25 | 25 | 25
pg/ml | 4 (2) | 5 (2) | -6 (2)

4. Secondary Outcome: Change in Plasma Insulin Concentration
Description: Measurement of change in plasma insulin concentration from baseline to 16 weeks following treatment with each study drug(s). Placebo arm was not included in this 16 week portion of the study, since subjects are diabetic. Only 3 arms of the study were conducted: (i) Byetta/Bydureon, (ii) Dapagliflozin (iii) Byetta/Bydureon plus Dapagliflozin.
Time Frame: Baseline to 16 weeks
Population: Type 2 diabetes
Measure: Mean (Standard Error); unit: microUnits/ml
Groups:
- Dapa+Exe: Therapy for 16 weeks with combination exenatide plus dapagliflozin
Arm/Group | Dapa+Exe | Dapa | Exenatide
Number analyzed (Participants) | 25 | 25 | 25
microUnits/ml | -2 (1) | -2 (2) | 3 (2)

5. Primary Outcome: Change in Endogenous Glucose Production (EGP) After 16 Weeks of Treatment With Each Study Drug.
Description: After screening, eligible subjects will receive a measurement of endogenous glucose production (EGP) with a prime-continuous infusion of 3-3H-glucose. The EGP measurement will be performed in the morning after a 10-12 hour overnight fast and will last 8.5 hours (from 6 AM to 2:30 PM). After a 3.5-hour tracer equilibration period, subjects (20 per group) will receive one of the following medications: (i) exenatide 5 ug subcutaneously; (ii) dapagliflozin (10 mg); and (iii) dapagliflozin 10 mg + exenatide 5 ug. Only three groups will be followed for 16 weeks since subjects are diabetic and placebo is not appropriate to use for this period. Again, subjects will be randomized to treatment with either exenatide, dapagliflozin or both drugs in combination. Repeat EGP will be measured again at 16 weeks as described above and data will be compared to respective "acute" studies.
Time Frame: 16 weeks
Population: Type 2 diabetes
Measure: Mean (Standard Error); unit: mg/kg.min
Groups:
- EXENATIDE: Exenatide:
  After 16 weeks of treatment with Exenatide, starting with 5 mcg twice daily and at 4 weeks changed to 2 mg once weekly subcutaneously.
- Dapagliflozin: After 16 weeks of treatment with Dapagliflozin, Farxiga, 10mg
- Exenatide Plus Dapagliflozin: After 16 weeks of therapy with both drugs in combination.
Arm/Group | EXENATIDE | Dapagliflozin | Exenatide Plus Dapagliflozin
Number analyzed (Participants) | 25 | 25 | 25
mg/kg.min | -0.23 (0.02) | 0.20 (0.03) | -0.12 (0.03)

ADVERSE EVENTS:
Time Frame: Baseline to 6 months
Description: Patient reporting and physical exam by principal investigator/nurse coordinator
Groups:
- Byetta / Bydureon: Exenatide:
  4 weeks of exenatide 5 mcg twice daily followed by Bydureon 2mg sc weekly
  Exenatide: Byetta 5 to 10 ug (twice daily) Bydureon 2mg (once weekly)
- Dapagliflozin: 16 weeks Dapagliflozin, Farxiga, 10mg
  Dapagliflozin: 10mg
- Byetta/Bydureon Plus Dapagliflozin: Exenatide:
  4 weeks of exenatide followed by 12 weeks of Bydureon 2mg sc once weekly PLUS
  Dapagliflozin:
  16 weeks Dapagliflozin, Farxiga, 10mg
  Dapagliflozin: 10mg
  Exenatide: Byetta 5 to 10 ug (twice daily) Bydureon 2mg (once weekly)
- Placebo: 16 weeks of placebo administration
Arm/Group | Byetta / Bydureon | Dapagliflozin | Byetta/Bydureon Plus Dapagliflozin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/15
Other Adverse Events (participants affected / at risk) | 6/25 | 4/25 | 7/25 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Byetta / Bydureon (N=25) | Dapagliflozin (N=25) | Byetta/Bydureon Plus Dapagliflozin (N=25) | Placebo (N=15)
Genital Mycosis (Reproductive system and breast disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0) — Nausea and Vomiting
Nausea and Vomiting (Gastrointestinal disorders) | 6 (6) | 0 (0) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT02981069/Prot_SAP_001.pdf